CLINICAL TRIAL: NCT07343804
Title: THE EFFECT OF ENDODONTIC TREATMENT ON CARDIOVASCULAR RISK BIOMARKERS IN PATIENTS WITH STABLE CORONARY ARTERY DISEASE : A RANDOMIZED CONTROLLED TRIAL
Brief Title: THE EFFECT OF ENDODONTIC TREATMENT ON CARDIOVASCULAR RISK BIOMARKERS IN PATIENTS WITH STABLE CORONARY ARTERY DISEASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nishant Chauhan
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Disease Risk Factor; Periapical Periodontitis
Keywords: cardiovascular disease; endodontic therapy; hs-CRP; IL-6
MeSH Terms: conditions — Periapical Periodontitis; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate treatment group (Experimental): Root canal will be done immediately after diagnosis of apical periodontitis.
  Interventions: Procedure: root canal treatment and intracanal medicament
- Delayed treatment group (Active Comparator): Root canal treatment will be done after 3 months
  Interventions: Procedure: root canal treatment and intracanal medicament

INTERVENTIONS:
Procedure: root canal treatment and intracanal medicament — Access opening will be done after rubber dam isolation and administration of local anesthesia. debridement of the pulp chamber will be done and all canal orifices will be identified. Negotiation of canals will be done. Working length will be determined using root ZX apex locator and will be verified radiographically. Coronal enlargement will be done using Gates-Glidden drills. The apical third of the root canal will be instrumented up to size 35 for mesial and up to size 45 for distal canals. Finally, root canals will be further instrumented with step-back technique enlargement in 1 mm increments to 3 sizes larger than the master apical file. Irrigation will be carried out using 5 mL of a 5% NaOCl solution between files. The root canals will be dried using paper points and filled with lateral condensed gutta-percha (Dentsply Maillefer) and Zinc oxide Eugenol based sealer mixed according to manufacturers' instructions.

SUMMARY:
Study subjects were obtained from the pool of OPD patients in the Department of Conservative Dentistry and Endodontics, PGIDS, Rohtak, and the Department of Cardiology, PGIMS, Rohtak. Baseline clinical, radiographic, and laboratory parameters (hsCRP and IL-6) were recorded. Patients were then randomly allocated to one of the two groups. In the test group, single-sitting root canal treatment was performed immediately, while in the control group, delayed endodontic intervention (after 3 months) was performed after three months. Clinical and laboratory parameters were again assessed at the end of 3 months in both groups. hsCRP and IL-6 indices were again done in the delayed treatment group after 3 months of root canal treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals 30 years of age and older, with a diagnosis of stable coronary artery disease (CAD) and chronic apical periodontitis.
2. All patients had to present with CAD defined by the Brazilian Society of Cardiology (Xavier et al., 2013) as the documented occurrence of one or more of the following events 6 months before entering the study: history of myocardial infarction, stable angina or ischaemia in non-invasive tests; surgical or percutaneous myocardial revascularization and lesion size of greater than 50% in at least one major coronary artery, as assessed by angiography; presence of angina and positive results of non-invasive testing of ischaemia.
3. Presence of apical periodontitis defined by the presence of at least 1 radiographic radiolucency ( ≥ 3mm) in teeth as assessed both clinically and radiographically ,with periapical index (PAI) scores ≥3 in a single permanent tooth and pulp necrosis verified by cold and electric pulp test.

   -

Exclusion Criteria:

1. Chronic conditions associated with periodontitis or with changes in systemic inflammation (e.g. diabetes mellitus, rheumatoid arthritis, rheumatic fever, malignancy, respiratory diseases, renal diseases).
2. Presence of localized or diffuse periodontal disease.
3. Acute symptomatic patients
4. Presence of CV risk factor - history of smoking
5. Acute conditions known to affect systemic inflammatory markers (orthopaedic trauma, surgery ,viral infections)
6. Medications (during last 3 months) known to affect systemic inflammatory markers (systemic steroids,immunosuppressants, hormone replacement therapy, contraceptives and systemic antibiotics
7. Obesity (body mass index [BMI]≥30 kg/m2
8. Pregnancy & Lactation.37

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the levels of hs-CRP and IL-6 in CAD patients with apical periodontitis. | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate institute of Dental Sciences, Rohtak, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No